CLINICAL TRIAL: NCT04396990
Title: A Randomized, Controlled, Masked (Reading Center) Prospective Study of the Effectiveness and Safety of the Ocular Therapeutix Dextenza 0.4 mg for the Treatment of Post-op. Inflammation and Pain in PRK
Brief Title: The RESTORE Study, A Randomized, Controlled, Masked (Reading Center) Prospective Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Tiffany Facile, Principal Investigator, Vance Thompson Vision
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: The RESTORE Study
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Refractive Surgery
MeSH Terms: interventions — Calcium Dobesilate; Prednisolone

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Dextenza (Experimental): Will receive Dextenza post-operative
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group B Topical Prednisolone (Active Comparator): Will receive standard of care prednisolone acetate 1% QID for 1 week, BID for 1 week
  Interventions: Drug: Topical Prednisolone

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion. The attributes of the insert reduce the risks for improper corticosteroid tapering and unwanted peaks and troughs in drug concentration.
  Arms: Group A Dextenza
Drug: Topical Prednisolone — Standard of care topical drop treatment
  Arms: Group B Topical Prednisolone

SUMMARY:
To determine patient preference and treatment outcomes with an intracanalicular dexamethasone (0.4mg) insert compared to standard steroid drop regimen in the contralateral eye following bilateral PRK surgery.

DETAILED DESCRIPTION:
Prospective Open-label Interventional Study Randomized, self-controlled design in which one eye (Group A) receives Dextenza and the second eye (Group B) receives prednisolone acetate 1% QID 1 week, BID 1 week following bilateral PRK surgery. All eyes will receive topical moxifloxacin QID for one week. Moxifloxacin in used post-op regardless of the research. Post-operative evaluations to be performed on Day 3 and Day 4, Month 1, and Month 3. Phone call survey to be performed on Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who is planned to undergo bilateral PRK surgery.
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Patients who are pregnant (must be ruled out in women of child-bearing age with pregnancy test).
* Active infectious ocular or systemic disease.
* Patients with active infectious ocular or extraocular disease.
* Patients actively treated with local or systemic immunosuppression including systemic corticosteroids.
* Patients with known hypersensitivity to Dexamethasone.
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator.
* Patients with a history of ocular inflammation or macular edema.
* Patients with allergy or inability to receive intracameral antibiotic.
* Patients on systemic non-steroidal anti-inflammatory drugs (NSAID) greater than 1,200 mg/day
* Patients with a corticosteroid implant (i.e. Ozurdex).
* Patient with corneal pathology which pre-disposes them to unsatisfactory outcomes.
* Patients who do not have 20/20 snellen visual acuity potential pre-operatively.
* MRSE greater than 6 diopters.
* Greater than 2 diopters anisometropia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Berdahl, MD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Group A Dextenza: Dextenza 0.4Mg Ophthalmic Insert Contralateral Eye Study
- Group B Topical Prednisolone: Topical Prednisolone: Standard of care topical drop treatment Contralateral Eye Study
Period: Overall Study
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Started | 20; 20 Eyes | 20; 20 Eyes
Completed | 20; 20 Eyes (Contralateral Eye Study. Each subject randomized to dextenza insert in one eye and topical steroid in contralateral eye.) | 20; 20 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- All Participants: 40 Eyes of 20 Patients.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [21 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Preference
Description: Primary outcome of patient reference of dexamethasone insert versus topical steroid as measured by adapted Comparison of Ophthalmic Medications for Tolerability (COMToL) questionnaire.
Time Frame: Through Month 1 (Day 28 +/- 3 days)
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: 40 Eyes of 20 Participants.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Participants
  Dexamethasone insert preference | 14
  Topical steroid preference | 4
  No preference | 2

2. Secondary Outcome: Percentage of Eyes Epithelialized at Day 3
Description: The percentage of eyes with fully healed epithelium at post-op day 3
Time Frame: Post-Operative Day 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- Dexamethasone Insert: 20 eyes that received dexamethasone insert
- Topical Steroid: 20 eyes that were treated with topical steroid
Arm/Group | Dexamethasone Insert | Topical Steroid
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
eyes
  Percent epithelialized at Day 3 | 20 | 20
  Percent not 100% epithelialized at Day 3 | 0 | 0

3. Secondary Outcome: Percentage of Eyes Fully Epithelialized at Day 4 Postoperative
Description: The percentage of eyes with fully healed epithelium at day 4 post-operative
Time Frame: Postoperative Day 4
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Insert | Topical Steroid
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
eyes
  Percentage of eyes fully epithelialized at day 4 | 19 | 20
  Percentage of eyes not fully epithelialized at day 4 | 1 | 0

4. Secondary Outcome: Mean Pain Score Per Eye (Group A: Dextenza vs. Group B: Topical Steroid)
Description: Pain score as measured by the Numerical Rating Scale (NRS) at day 3 post-operative. The rating scale is from 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dextenza Group Pain Score: Pain score at Postoperative Day 3 for Dextenza group
- Topical Steroid Group Pain Score: Pain score at Postoperative Day 4 for Topical steroid group
Arm/Group | Dextenza Group Pain Score | Topical Steroid Group Pain Score
Number analyzed (Participants) | 20 | 20
score on a scale | 0.9 (0.995) | 0.850 (0.853)

5. Secondary Outcome: SPEED Questionnaire Results at Baseline and Postoperative Day 28
Description: Patient evaluation of eye dryness measured by a modified SPEED questionnaire with a results recorded 0-28 with 28 being the most severe.
Time Frame: Pre-op Visit and Month 1 (Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dexamethasone Insert Group: Eyes inserted with dexamethasone insert
- Topical Steroid Group: Eyes treated with topical steroid
Arm/Group | Dexamethasone Insert Group | Topical Steroid Group
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 3.75 (4.05) | 3.70 (4.11)
  Day 28 | 4.00 (4.07) | 4.22 (4.98)

6. Secondary Outcome: Uncorrected Distance Visual Acuity
Description: measured using the ETDRS acuity chart at 4 meters recorded in logMAR.
Time Frame: Month 1 and Month 3.
Population: A total of 40 eyes of 20 participants was analyzed
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Dexamethasone Insert Group; Topical Steroid Group: Uncorrected distance visual acuity
Arm/Group | Dexamethasone Insert Group | Topical Steroid Group
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 20 | 20
logMAR
  Uncorrected distance visual acuity at month 1 | 0.0005 (0.121) | -0.073 (0.067)
  Uncorrected distance visual acuity at month 3 | -1.117 (0.068) | -0.153 (0.057)

7. Secondary Outcome: Spectacle Corrected Distance Visual Acuity at Months 1 and 3 Post-operative
Description: Best-corrected distance visual acuity measured using ETDRS acuity chart at 4 meters, recorded in logMAR notation
Time Frame: Month 1 and Month 3
Population: 40 eyes of 20 participants analyzed
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Dexamethasone Insert Arm; Topical Steroid Arm: Corrected distance visual acuity measured at postoperative month 1 and month 3
Arm/Group | Dexamethasone Insert Arm | Topical Steroid Arm
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
logMAR
  Month 1 | -0.051 (0.066) | -0.093 (0.050)
  Month 3 | -0.146 (0.043) | -0.167 (0.044)

ADVERSE EVENTS:
Time Frame: Data collected through 3 months.
Groups:
- Dexamethasone Insert Arm: Eyes implanted with dexamethasone insert
- Topical Steroid Arm: Eyes implanted with topical steroid
Arm/Group | Dexamethasone Insert Arm | Topical Steroid Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT04396990/Prot_001.pdf
  • Informed Consent Form (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT04396990/ICF_002.pdf